CLINICAL TRIAL: NCT05376267
Title: Pediatric Influence of Cooling Duration on Efficacy in Cardiac Arrest Patients (P-ICECAP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Kennedy Krieger Institute, Baltimore, MD (Unknown)
Responsible Party: Principal Investigator, Frank W. Moler, M.D, M.S, Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDE G210126; 1UG3HL159134-01 (NIH); U24HL159132 (NIH); HUM00206424 (Other: UM IRB NUMBER)
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Hypothermia, Induced; Hypoxia-Ischemia, Brain
Keywords: Bayesian Adaptive Clinical Trial; Hypothermia, therapeutic; Coma; Pediatric
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypothermia; Hypoxia-Ischemia, Brain; Coma | interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: Bayesian Adaptive Design
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blinded to the treatment assignment of the participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (10):
- Cooling 0 hours (Experimental): Participants will be kept at a normal temperature for the whole 5 days.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 12 hours (Experimental): The participant will be cooled to 33°Celsius (C) for 12 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 18 hours (Experimental): The participant will be cooled to 33°C for 18 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 24 hours (Experimental): The participant will be cooled to 33°C for 24 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 36 hours (Experimental): The participant will be cooled to 33°C for 36 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 48 hours (Experimental): The participant will be cooled to 33°C for 48 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 60 hours (Experimental): The participant will be cooled to 33°C for 60 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 72 hours (Experimental): The participant will be cooled to 33°C for 72 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 84 hours (Experimental): The participant will be cooled to 33°C for 84 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia
- Cooling 96 hours (Experimental): The participant will be cooled to 33°C for 96 hours, slowly rewarmed over approximately 16 hours, and then will be kept at a normal temperature (36.8°C or 98.6°F) until the end of the 5th day.
  Interventions: Device: Therapeutic Hypothermia

INTERVENTIONS:
Device: Therapeutic Hypothermia — Participants will receive therapeutic hypothermia for the assigned number of hours with controlled rewarming,
  A zero hour cooling duration (normothermia) treatment arm will be opened for enrollment if there is not an increase in the treatment effect across the durations. Alternatively, longer durations (84 or 96 hours) will be opened for enrollment if the treatment effects are increasing (rather than plateauing or decreasing) through 72 hours.

SUMMARY:
This is a multicenter trial to establish the efficacy of cooling and the optimal duration of induced hypothermia for neuroprotection in pediatric comatose survivors of cardiac arrest.

The study team hypothesizes that longer durations of cooling may improve either the proportion of children that attain a good neurobehavioral recovery or may result in better recovery among the proportion already categorized as having a good outcome.

ELIGIBILITY:
Inclusion criteria:

* Age 2 days to < 18 years with corrected gestational age of at least 38 weeks
* Chest compressions for at least 2 minutes
* Coma or encephalopathy after resuscitation from Out-of-Hospital Cardiac Arrest (OHCA)
* Requires continuous mechanical ventilation through endotracheal tube or tracheostomy
* Definitive temperature control device initiated
* Randomization within 6 hours of Return of Spontaneous Circulation (ROSC)
* Informed consent from Legally Authorized Representative (LAR) including intent to maintain life support for 120 hours

Exclusion criteria:

* Glasgow Coma Motor Score (GCMS) = 6
* LAR does not speak English or Spanish
* Duration of Cardiopulmonary Resuscitation (CPR) > 60 minutes
* Severe hemodynamic instability with continuous infusion of epinephrine or norepinephrine of 2 micrograms per kilogram per minute (μg/kg/minute) or initiation of Extracorporeal membrane oxygenation (ECMO)
* Pre-existing severe neurodevelopmental deficits with Pediatric Cerebral Performance Category (PCPC) =5 or progressive degenerative encephalopathy
* Pre-existing terminal illness, unlikely to survive to one year
* Cardiac arrest associated with brain, thoracic, or abdominal trauma
* Active and refractory severe bleeding prior to randomization
* Extensive burns or skin lesions incompatible with surface cooling
* Planned early withdrawal of life support before 120 hours
* Sickle cell anemia
* Pre-existing cryoglobulinemia
* Non-fatal drowning in ice covered water
* Central nervous system tumor with ongoing chemotherapy
* Previous enrollment in P-ICECAP trial
* Prisoner
* Chronic hypothermia
* New post-cardiac arrest diabetes insipidus
* Pregnancy

Ages: 2 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales - Third Edition (VABS-3) Mortality Composite Score at 12 months after return of spontaneous circulation | 12 months after out-of-hospital cardiac arrest
  The VABS-3 score, designed to be administered to surviving children with any level of function including comatose status to age-appropriate neurobehavioral functioning, ranges from 20 to 140 with age-corrected standardized mean and standard deviation of 100 and 15, respectively. Deaths will be scored as 0 in this trial.

SECONDARY OUTCOMES:
Change in Pediatric Cerebral Performance Category (PCPC) at 12 months from baseline | Baseline and 12 months after cardiac arrest
  The Pediatric Cerebral Performance Category is a global scale based on observer impressions. It's a six point graded scale of increasing disability from 1 normal function, to 6 death. Scores include 1 for good, 2 for mild disability, 3 for moderate disability, 4 for severe disability, and 5 for vegetative state or coma. Higher scores indicating worse performance or functional morbidity.
Pediatric Resuscitation after Cardiac Arrest (PRCA) at 12 months | 12 months after cardiac arrest
  The PRCA adapted from the Pediatric Stroke Outcome measure, ranges from 0-21 where lower scores indicate less impairment. Deaths will be assigned the worst score of 21 for PRCA.
Survival at 12 months | 12 months after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Frank Moler, MD, Principal Investigator — University of Michigan; Alex Topjian, MD, Principal Investigator — Children's Hospital of Philadelphia; William Meurer, MD, Principal Investigator — University of Michigan
Locations (56):
- United States (46):
  - University of Alabama at Birmingham / Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Memorial Health - Miller Children's and Women's Hospital of Long Beach, Long Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California Los Angeles (UCLA) Mattel Children's Hospital, Los Angeles, California
  - University of California - Oakland / UCSF Benoiff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, Davis, Sacramento, California
  - University of California - San Francisco (UCSF) Benioff Children's Hospital San Francisco, San Francisco, California
  - Stanford, Santa Clara, California
  - University of Florida (UF) Health Shands Children's Hospital, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, University of Chicago, Chicago, Illinois
  - Children's Hospital of Illinois, Peoria, Illinois
  - Riley Children's Health, Indianapolis, Indiana
  - University of Iowa, Carver College of Medicine, Iowa City, Iowa
  - University of Maryland Children's Hospital, Baltimore, Maryland
  - Johns Hopkins Medicine Children's Center, Baltimore, Maryland
  - MassGeneral Hospital for Children, Boston, Massachusetts
  - University of Michigan CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Fairview Masonic Children's Hospital, Minneapolis, Minnesota
  - Washington University / St. Louis Children's Hospital, St Louis, Missouri
  - University of Buffalo / Oishei Children's Hospital, Buffalo, New York
  - Cohen Children's Medical Center of NY / Northwell Health, New Hyde Park, New York
  - Mount Sinai Icahn / Kravis Children's Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University / Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oregon Health & Science University Doernbecher Children's Hospital, Portland, Oregon
  - Penn State University / Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh (UPMC), Pittsburgh, Pennsylvania
  - University of Tennesses Health Center / Le Bonheur Children's, Memphis, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - Texas Children's Hospital, Baylor, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, University of Utah School of Medicine, Salt Lake City, Utah
  - American Family Children's Hospital, Madison, Wisconsin
  - Children's Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Queensland Children's Hospital, Brisbane, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- Birmingham Children's Hospital, United Kingdom, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in the NHLBI data repository after trial completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after publication on main outcome results paper
Access Criteria: Data use agreement with the appropriate NHLBI repository

DOCUMENTS (2):
  • Study Protocol (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT05376267/Prot_000.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT05376267/ICF_001.pdf